CLINICAL TRIAL: NCT03025217
Title: Total Lifestyle Coaching Pilot Study (TLC)
Acronym: TLC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Michelle Dossett, MD, PhD, MPH, Assistant Physician, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014P001549
Record Dates: First submitted 2017-01-17; First posted 2017-01-19 (Estimated); Results first posted 2019-02-20 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Obesity; Weight Loss; Telemedicine
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TLC Program (Experimental): The TLC Program consists of one in-person visit with a licensed dietician and biweekly phone coaching sessions. During the program, the dietician will 1) identify specific nutrition goals, 2) review and tailor the education materials to the patient's needs, and 3) set up regular telephone coaching sessions of up to two sessions per month for six months for each patient. Motivational interviewing and nutrition/health coaching will be provided.
  Interventions: Behavioral: Total Lifestyle Coaching (TLC)

INTERVENTIONS:
Behavioral: Total Lifestyle Coaching (TLC)

SUMMARY:
The investigators aim to develop, pilot and evaluate a new "Total Lifestyle Coaching" (TLC) program, that will address both information and behavior-change aspects of nutrition education for patients whose body mass index (BMI) exceeds 25.

DETAILED DESCRIPTION:
This is a single-arm pilot study of patients at the Revere Healthcare Center with a BMI greater than 25. The intervention consists of a single in-person assessment with a dietician followed by telephone coaching sessions addressing nutrition, sleep, stress-reduction skills, and physical activity over the course of 6 months. Study team assessed anthropomorphic, demographic, and behavioral measures prior to the initial dietician assessment and at study completion (6 months following enrollment). Semi-structured exit interviews assessing participants' experiences in the program were also conducted following program completion.

ELIGIBILITY:
Inclusion Criteria:

1. age 21 and older
2. body mass index (BMI) exceeds 25
3. speaks English
4. has access to a telephone
5. able to come into MGH-Revere health center for at least four face-to-face meetings over a six month period.
6. overweight (BMI exceeds 25)

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-09; Primary Completion 2015-08 (Actual); Study Completion 2016-11 (Actual)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chad-Friedman E, Pearsall M, Miller KM, Wheeler AE, Denninger JW, Mehta DH, Dossett ML. Total Lifestyle Coaching: A Pilot Study Evaluating the Effectiveness of a Mind-Body and Nutrition Telephone Coaching Program for Obese Adults at a Community Health Center. Glob Adv Health Med. 2018 Jul 4;7:2164956118784902. doi: 10.1177/2164956118784902. eCollection 2018. PMID 30013821

RESULTS

PARTICIPANT FLOW:
Groups:
- TLC Program: The TLC Program consists of one in-person visit with a licensed dietician and biweekly phone coaching sessions. During the program, the dietician will 1) identify specific nutrition goals, 2) review and tailor the education materials to the patient's needs, and 3) set up regular telephone coaching sessions of up to two sessions per month for six months for each patient. Motivational interviewing and nutrition/health coaching will be provided.
  Total Lifestyle Coaching (TLC)
Period: Overall Study
Arm/Group | TLC Program
Started | 31
Completed | 27
Not Completed | 4
Not completed — Pregnancy | 1
Not completed — Lost to Follow-up | 1
Not completed — Not eligible, poor English | 2

BASELINE CHARACTERISTICS:
Arm/Group | TLC Program
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 23
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight
Description: Change in weight between baseline (week 0) and post intervention (week 26)
Time Frame: 26 weeks
Population: Program Completers
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | TLC Program
Number analyzed (Participants) | 27
pounds
  Baseline | 209 (35.5)
  26 weeks | 205 (36.7)
Statistical Analysis 1: Comparison: TLC Program; Test type: Other; p = .095, t-test, 2 sided; Cohen's d = 0.33

2. Secondary Outcome: Perceived Stress Scale
Description: Change in perceived stress as measured by the PSS-10 questionnaire administered at baseline (week 0) and post intervention (week 26). Score range is 0 - 40 with higher scores indicating higher perceived stress.
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TLC Program
Number analyzed (Participants) | 27
score on a scale
  Baseline | 19 (7.1)
  26 weeks | 13 (7.5)
Statistical Analysis 1: Comparison: TLC Program; Test type: Other; p = .001, t-test, 2 sided; Cohen's d = 0.75

ADVERSE EVENTS:
Arm/Group | TLC Program
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes